CLINICAL TRIAL: NCT02253407
Title: A Phase IV, Non-Inferiority, Observer Blind Randomized Clinical Study Comparing Safety And Immunogenicity Of MMR Subcutaneous Vaccination By Disposable-Syringe Jet Injector To Vaccination By Needle And Syringe For The Administration In Healthy Children In India Aged 15 To 18 Months
Brief Title: Safety & Immunogenicity of MMR Vaccine by DSJI to That by Needle-Syringe in 15-18 Months Old Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Serum Institute of India Pvt. Ltd. (Industry)
Collaborators: PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MMR-01/12; CTRI/2013/05/003702 (Registry Identifier: Clinical Trial Registry of India)
Record Dates: First submitted 2014-09-27; First posted 2014-10-01 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Immune Response to MMR Vaccine
MeSH Terms: interventions — Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Disposable syringe jet injector (Experimental): Subjects in this arm will be given a single subcutaneous 0.5 mL dose of Serum Institute of India Ltd.'s MMR vaccine (Brand name: Tresivac) via Disposable Syringe Jet Injector (Brand Name:Stratis) of Pharmajet Inc.
  Interventions: Biological: MMR vaccine
- Needle-Syringe (Active Comparator): Subjects in this arm will be given a single subcutaneous 0.5 mL dose of Serum Institute of India Ltd.'s MMR vaccine (Brand name: Tresivac) via conventional needle and Syringe
  Interventions: Biological: MMR vaccine

INTERVENTIONS:
Biological: MMR vaccine
  Other Names: Tresivac

SUMMARY:
This is a study planned to determine and compare immunogenicity and reactogenicity of MMR vaccine of SIIL delivered either with disposable-Syringe Jet Injector (DSJI) or disposable-syringe needle in total 340 Indian infants aged 15 to 18 months.

DETAILED DESCRIPTION:
This is a randomized, observer blind, non-inferior, parallel group, multi-centre clinical study to determine and compare immunogenicity and reactogenicity of MMR vaccine of SIIL delivered either with disposable-Syringe Jet Injector (DSJI) or disposable-syringe needle in total 340 Indian infants aged 15 to 18 months. Sera samples will be analyzed by ELISA for seroconversion / seropositivity for each individual component of vaccine i.e. measles, mumps and rubella at 35 days after administration of a single dose of MMR vaccine of Serum Institute of India.

ELIGIBILITY:
Inclusion Criteria:

1. Normal healthy infants of age 15-18 months at the time of the screening and have not received their first dose of MMR vaccine.
2. Previously received a measles monovalent vaccine at 9 months, as confirmed by the childhood vaccination record.
3. Parents or legal guardians of subject willing to give written informed consent and willing to comply with study protocol.
4. Free of obvious health problems as established by medical history and screening evaluation including clinical examination.

Exclusion Criteria:

1. Infant subject participating in other clinical trial or planned participation in another clinical trial during the present trial period
2. Infant with congenital or acquired immunodeficiency, malignancy or receiving immunosuppressive therapy.
3. Infant with history of allergy or systemic hypersensitivity to any of the vaccine component or to a vaccine containing the same substances.
4. Infant with history of epilepsy or a seizure disorder or neurodevelopmental disorders.
5. Clinical history of measles, mumps, or rubella infection.
6. Infants with leukemia, lymphoma, or any other cancer or neoplasm.
7. Acute or chronic, clinically significant pulmonary, endocrine, autoimmune, neurological, cardiovascular, metabolic, hepatic or renal functional abnormality, as determined by medical history, and physical examination tests, which in the opinion of the investigator, might interfere with the study objectives
8. Infant with any other condition, which, in the opinion of the investigator would jeopardize the safety or rights of the infant participating in the study or making it unlikely the subject could complete the protocol.

Ages: 15 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 341 (Actual)
Dates: Start 2014-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Seropositivity of individual child for measles, mumps and rubella | 35 days after administration of the study vaccines
  Seropositivity of the individual child for particular vaccine component will be defined according to the levels given in the kit literature.

SECONDARY OUTCOMES:
Comparison of Geometric Mean titers (GMTs) for anti-measles, anti-mumps and anti-rubella antibodies | Day 35
Solicited adverse reactions | Day 14
Unsolicited adverse events | Day 35
Serious adverse events (SAEs) | Day 35

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Bavdekar, MD, Principal Investigator — Department of Pediatrics, KEM Hospital Research Centre, Pune, India; Jitendra Oswal, MD, Principal Investigator — Department of Pediatrics, Bharati Vidyapeeth Deemed University Medical College and Hospital, Pune, India
Locations (6):
- India (6):
  - Department of Paediatrics, Andhra Medical College, King George Hospital, Maharanipet,, Visakhapatnam, Andhra Pradesh
  - Krishna Institute of Medical Sciences Deemed University,, Karad, Maharashtra
  - Shirdi Sai Baba Rural Hospital, KEM Hospital Research Centre, Vadu Rural Health Program, Vadu Budruk, Tal: Shirur, Pune, Maharashtra
  - Department of Pediatrics, KEM Hospital Research Centre, Sardar Moodliar Road, Rasta Peth,, Pune, Maharashtr
  - Department of Pediatrics, Bharati Vidyapeeth Deemed University Medical College and Hospital, Satara Road, Katraj, Dhankawadi, Pune, Maharasthra
  - Dept of Pediatrics, Sri Ramachandra Medical Centre, No. 1, Ramachandra nagar, Porur,, Chennai, Tamil Nadu

REFERENCES:
- [Result] Bavdekar A, Oswal J, Ramanan PV, Aundhkar C, Venugopal P, Kapse D, Miller T, McGray S, Zehrung D, Kulkarni PS; SII MMR author group. Immunogenicity and safety of measles-mumps-rubella vaccine delivered by disposable-syringe jet injector in India: A randomized, parallel group, non-inferiority trial. Vaccine. 2018 Feb 21;36(9):1220-1226. doi: 10.1016/j.vaccine.2018.01.006. Epub 2018 Feb 1. PMID 29395526